CLINICAL TRIAL: NCT03545256
Title: Open Non-randomized Study on the Management of Operable T1-N0 or T2-N0 Oral Cavity and Oropharynx Cancer and Sentinel Lymph Node in Outpatient Surgery
Brief Title: Sentinel. Ambulatory. Oral Cavity. Oropharynx (S.A.C.O)
Acronym: SACO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL17_0165
Record Dates: First submitted 2018-05-07; First posted 2018-06-04 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cancer T1-N0 or T2-N0 of the Oral Cavity
Keywords: Outpatient; head neck cancer; Lymph node metastasis; surgery; Quality of life; economical study
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphatic Metastasis | interventions — Ambulatory Surgical Procedures

STUDY DESIGN:
Intervention Model Description: The surgical procedure associated with the sentinel lymph node technique is carried out in two stages:
  - Lymphoscintigraphy at Day-1 : This is the identification of the lymphatic network of the patient by a prior injection of radioactive tracer, nanocolloide labeled with technetium99, around the primary tumor.
  - Surgery on D0: The patient is admitted to the hospital at 7:00 am in outpatient unit. He is reviewed by the anesthetist before the intervention and is transferred to the operating room for the intervention under AG.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- T1-N0 or T2-N0 cancers of the oral cavity (Other): outpatient surgery for T1-N0 or T2-N0 cancers of the oral cavity or oropharynx with lymph node search
  Interventions: Procedure: outpatient surgery for T1-N0 or T2-N0 cancers of the oral cavity or oropharynx with lymph node search

INTERVENTIONS:
Procedure: outpatient surgery for T1-N0 or T2-N0 cancers of the oral cavity or oropharynx with lymph node search — The surgical procedure associated with the sentinel lymph node technique is carried out in two stages:
  - Lymphoscintigraphy at Day-1 : This is the identification of the lymphatic network of the patient by a prior injection of radioactive tracer, nanocolloids labeled with technetium99, around the primary tumor. A planar CT image acquisition is performed to identify the sentinel lymph nodes (Gs(s)) which are then marked on the skin with an indelible marker.
  Surgery on D0:
  The patient is admitted to the hospital at 7:00 am in outpatient unit. He is reviewed by the anesthetist before the intervention and is transferred to the operating room for the intervention under AG.
  The main tumor is operated by mouth.

SUMMARY:
This is a single-center pilot study of open-label, non-randomized interventional research based on the outpatient management of 30 patients with T1-N0 or T2-N0 cancer in the oral cavity or oropharynx.

DETAILED DESCRIPTION:
Currently, patients with oral cancer or oropharynx T1-N0 or T2-N0 are treated by surgery on the tumor and the neck, both validated techniques are either with a systematic lymph node dissection or a search for lymph sentinel node (GS). The goal on the lymph sentinel nodes is to diagnose the presence of metastasis (s). With the GS technique, the length of hospital stay can be shorter. The limited invasiveness of tumor surgery of the oral cavity and oropharynx and GS and short postoperative monitoring is compatible with outpatient management, so it should be evaluated through a study clinical.

The main objective of this study is to evaluate the rate of conversion to complete hospitalization or re-hospitalization within 10 days of surgery J0. The secondary objectives are the evaluation of the acceptance rate of outpatient surgery by the eligible patient, complications related to outpatient management, the quality of life of the patient and the cost of the strategy over the first month following J0.

The surgical procedure associated with the sentinel lymph node technique is carried out in two stages:

- Lymphoscintigraphy at Day-1 : This is the identification of the lymphatic network of the patient by a prior injection of radioactive tracer, nanocolloids labeled with technetium99, around the primary tumor. A planar or 3-minute CT image acquisition is performed 30 to 60 minutes after injection in anteroposterior and lateral view to identify the sentinel lymph nodes (GS(s)) which are then marked on the skin with an indelible marker. This routine care examination is done in an external act.

- Surgery on D0: The patient is admitted to the hospital at 7:00 am in outpatient unit. He is reviewed by the anesthetist before the intervention and is transferred to the operating room for the intervention under General anesthesia.

The main tumor is operated by mouth. The ganglionic surgical procedure consists of the removal of the GS(s) by a limited cervical approach, following a cervical dissection line. The GS(s) are identified by a gamma detection probe, equipped with a high-resolution collimator whose tip is covered with a sterile disposable sleeve. Exeresis of the GS(s) is performed by removing the peri-ganglionic cellular tissue and avoiding any capsular intrusion. The GS lymph node (s) so taken is sent freshly by special request to the pathologist for final analysis according to the recommended procedure for GS.

The cervical dissection will be performed later if the definitive analysis finds a ganglionic invasion. In this case, the patient will be re-hospitalized in unit full hospitalization for cervical lymph node dissection: the ganglionic areas systematically concerned are the levels I, II, III and IV for tumors of the oral cavity and II, III and IV for the oropharynx. The gesture will be bilateral if the lymphoscintigraphy had found a bilateral drains. The cervical dissection parts are labeled and sent for routine final pathological analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old with no upper age limit
* Patient (s) affiliated to a social security system, or beneficiary of such a system
* Patient information and informed consent signed by the patient
* Patient no longer participating in another trial since legal time
* Patient with primary squamous cell carcinoma of the oral cavity or oropharynx documented by biopsy with histological analysis less than 1 month old
* Tumor operable by TNM stage, location and general condition of the patient
* Systematic Oto-Rhino-Laryngology panendoscopy eliminating a second synchronous tumor and establishing precisely the T
* Stage T1 or T2, N0 and M0
* Proposal by a multidisciplinary meeting for tumor surgery and GS technique
* Eligibility criteria for ambulatory surgery present
* Anesthetic criteria for eligibility for outpatient hospitalization (ref AFAR 29 (2010) 67-72, formalized expert recommendations) including ASA I, II and III score stable
* Patient able to understand the nature, purpose and methodology of the study

Exclusion Criteria:

* lack of one of the inclusion criteria
* other cancer being treated
* non-infiltrating tumor: high grade dysplasia, carcinoma in situ
* insufficient tumor excision: invaded margins without complementary recovery in healthy zone
* contraindication to sentinel lymph node surgery or ganglion dissection
* contraindication to radiotherapy
* contraindications to performing a scintigraphy:
* Known allergy or intolerance to the injected product and in particular to Technetium-99
* Pregnancy
* Refusal to accept the entire treatment (nodal diagnosis on GS, lymph node dissection pN + follow-up of adjuvant radiotherapy if necessary)
* impossible to follow over 2 years
* refusal to accept the monitoring described and / or to provide the information necessary for the study
* patient already treated for this tumor outside of an excisional biopsy
* patient who previously had chemotherapy or immunotherapy for another cancer outside the VADS in a period of less than 6 months
* patient who has had cervical or VADS radiotherapy regardless of the cause or delay
* patient who has had previous cervical surgery regardless of cause or delay
* Patient protected by law (patient under guardianship).
* Patient (e) deprived of liberty by administrative decision.
* Pregnant or lactating women according to article L1121-5 of the CSP. An assay of βHCG will be performed routinely to ensure the absence of pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Conversion rate in complete hospitalization or re-hospitalization within 10 days following the surgical procedure (D0) | From Day 0 to 10 days post surgery
  the conversion into complete hospitalization on the day of the procedure (Day 0) or re-hospitalization within 10 days following the surgical procedure (Day 0) respectively will be performed in case of medical or surgical complications or according to the doctor's opinion for the release of the patient, or in case of lymph nodes dissection

SECONDARY OUTCOMES:
Acceptance rate of outpatient surgery | inclusion visit
  Acceptance rate of outpatient surgery validated by the multidisciplinary meeting and proposed to the patient who meets the eligibility criteria for the inclusion visit
Description of complications attributable to outpatient care taken on Day 0, Day 10 and Month1 | From Day 0 to Month 1 post surgery
  All complications related to outpatient care will be recorded
Quality of life at inclusion visit | Inclusion visit
  self-questionnaire completed by the patient at inclusion visit, Score reported by the subjects on the Quality of life questionnaire QLQ-C30. The scores of the different scales are between 0 and 100. A score of the overall health of quality of life (QoL) close to 100 indicates a QoL close to perfect health. Similarly, a score of a functional scale close to 100 represents a level close to perfect capacity.
Quality of life at Day 0 visit | Day 0 visit
  self-questionnaire completed by the patient at visit Day 0 visit, Scores reported by the subjects on the Quality of life questionnaires QLQ-H & N35.
  The questionnaire EORTC QLQ- H & N35 contains 35 questions that incorporate 7 multidimensional scales that assess pain, swallowing, senses (taste and smell), speech, socializing, social contacts, and sexuality during the previous week. It also includes 11 isolated items.
  The scoring approach for the QLQ-H & N35 questionnaire is identical in principle to that of the QLQC30 questionnaire symptom scales.
Quality of life at Day 10 post surgery | Day 10 visit post surgery
  self-questionnaire completed by the patient at visit Day 10 visit, Scores reported by the subjects on the Quality of life questionnaires QLQ-H & N35.
  The questionnaire EORTC QLQ- H & N35 contains 35 questions that incorporate 7 multidimensional scales that assess pain, swallowing, senses (taste and smell), speech, socializing, social contacts, and sexuality during the previous week. It also includes 11 isolated items.
  The scoring approach for the QLQ-H & N35 questionnaire is identical in principle to that of the QLQC30 questionnaire symptom scales.
Quality of life at month 1 post surgery | Month 1 visit post surgery
  self-questionnaire completed by the patient at inclusion Month 1 visit. Scores reported by the subjects on the Quality of life questionnaire SF-36.Score from the worst health condition imaginable (0) to the best state of health imaginable (100).
Evaluation of the cost of the strategy at Month 1 | Month 1
  Description: The cost will be evaluated on the first month of outpatient management

CONTACTS AND LOCATIONS:
Overall Officials: Renaud GARREL, ENT, Principal Investigator — CHU Montpellier Gui de Chauliac Hospital, Neuroscience Head and Neck Pole, ENT Department
Locations (1):
- Gui de Chauliac Hospital, ENT Department 80 rue Augustin Fliche, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burcia V, Costes V, Faillie JL, Gardiner Q, de Verbizier D, Cartier C, Jouzdani E, Crampette L, Guerrier B, Garrel R. Neck restaging with sentinel node biopsy in T1-T2N0 oral and oropharyngeal cancer: Why and how? Otolaryngol Head Neck Surg. 2010 Apr;142(4):592-7.e1. doi: 10.1016/j.otohns.2009.12.016. PMID 20304284
- [Background] Garrel R, Poissonnet G, Temam S, Dolivet G, Fakhry N, de Raucourt D. Review of sentinel node procedure in cN0 head and neck squamous cell carcinomas. Guidelines from the French evaluation cooperative subgroup of GETTEC. Eur Ann Otorhinolaryngol Head Neck Dis. 2017 Apr;134(2):89-93. doi: 10.1016/j.anorl.2016.10.004. Epub 2016 Nov 11. PMID 27842990
- [Background] Schilling C, Stoeckli SJ, Haerle SK, Broglie MA, Huber GF, Sorensen JA, Bakholdt V, Krogdahl A, von Buchwald C, Bilde A, Sebbesen LR, Odell E, Gurney B, O'Doherty M, de Bree R, Bloemena E, Flach GB, Villarreal PM, Fresno Forcelledo MF, Junquera Gutierrez LM, Amezaga JA, Barbier L, Santamaria-Zuazua J, Moreira A, Jacome M, Vigili MG, Rahimi S, Tartaglione G, Lawson G, Nollevaux MC, Grandi C, Donner D, Bragantini E, Dequanter D, Lothaire P, Poli T, Silini EM, Sesenna E, Dolivet G, Mastronicola R, Leroux A, Sassoon I, Sloan P, McGurk M. Sentinel European Node Trial (SENT): 3-year results of sentinel node biopsy in oral cancer. Eur J Cancer. 2015 Dec;51(18):2777-84. doi: 10.1016/j.ejca.2015.08.023. Epub 2015 Nov 18. PMID 26597442
- [Background] Lee MK, Nalliah RP, Kim MK, Elangovan S, Allareddy V, Kumar-Gajendrareddy P, Allareddy V. Prevalence and impact of complications on outcomes in patients hospitalized for oral and oropharyngeal cancer treatment. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Nov;112(5):581-91. doi: 10.1016/j.tripleo.2011.06.032. PMID 22035652